CLINICAL TRIAL: NCT07268235
Title: Timing of Oocyte Retrieval and Micro Testicular Sperm Extraction: Does it Make a Difference? A Single-center Retrospective Cohort
Brief Title: Timing of Oocyte Retrieval and Micro Testicular Sperm Extraction
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: Micro-TESE
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Microdissection Testicular Sperm Extraction
Keywords: Nonobstructive Azoospermia; oligoasthenoteratozoospermia; intracytoplasmic sperm injection; In vitro fertilization; cryptozoospermia
MeSH Terms: conditions — Azoospermia, Nonobstructive; Oligospermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective study to assess outcomes of micro-TESE performed 24 or 48 hours before oocyte retrieval and ICSI.

DETAILED DESCRIPTION:
This retrospective study evaluates patients undergoing ICSI following micro-TESE. Participants are assigned to two groups based on the interval between sperm extraction and oocyte retrieval (24 vs. 48 hours). Clinical and embryological outcomes from the first embryo transfer will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men who underwent a micro-TESE at the OVO clinic from June 2015 to January 2025.
* Patients with non-obstructive azoospermia (NOA), (absence of spermatozoa in multiple semen analyses)
* Patients with cryptozoospermia, (presence of a small number of spermatozoa detectable only after semen centrifugation)
* Patients with oligoasthenoteratozoospermia (OAT), (sperm concentration of less than 15 million/mL, reduced motility and abnormal morphology)

Exclusion Criteria:

* Patients who did not have any sperm noted following micro-TESE
* Use of donor sperm or oocytes
* Frozen sperm or oocytes
* Same day oocyte retrieval and sperm extraction
* Reversible cause of cryptozoospermia (i.e presence of a varicocele, febrile illness, or recent toxin exposure) Partial genital tract obstruction (i.e post-vaso-vasostomy, post-vasoepididymostomy, and low volume cryptozoospermia with ejaculatory duct obstruction)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men who underwent a micro-TESE for IVF treatment
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2025-11-15 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Number of live births following ICSI with micro-TESE either 24 or 48 hours prior to oocyte retrieval | For IVF performed from June 2015 to January 2025

SECONDARY OUTCOMES:
Percentage of fertilized oocytes with two pronuclei (2PN) | For IVF performed from June 2015 to January 2025
Percentage of usable blastocyst (defined as frozen and transferred blastocysts) | For IVF performed from June 2015 to January 2025
Pregnancy rate based on positive β-hCG | For IVF performed from June 2015 to January 2025

CONTACTS AND LOCATIONS:
Overall Officials: Isaac-Jacques Kadoch, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No